CLINICAL TRIAL: NCT01134120
Title: A Phase 1 Study of LY2784544 in Patients With JAK2 V617F-Positive Myeloproliferative Disorders
Brief Title: A Study in Myeloproliferative Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13201; I3X-MC-JHTA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — LY2784544

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2784544 (Experimental)
  Interventions: Drug: LY2784544

INTERVENTIONS:
Drug: LY2784544 — LY2784544 will be supplied as a capsule. The study drug will be taken by mouth daily while the patient is on study. In this study, different patients will be treated at different doses of LY2784544 until reaching the highest dose that patients can tolerate.

SUMMARY:
The purpose of this study is to find out the safe dose range of the study drug in patients with myeloproliferative disorders.

DETAILED DESCRIPTION:
The purpose of the study is to learn:

1. How much and how often LY2784544 should be given to patients
2. What is the safety profile of LY2784544 and any side effects that might be associated with it
3. How LY2784544 is taken up, distributed, broken down, and passed out of your body
4. Whether LY2784544 can help patients with myeloproliferative disorders
5. If any markers in the blood (biomarkers) can identify patients who will respond better to the study drug.

The planned duration of the study is not fixed. The length of time patients participate in the study will be determined by the investigator/study doctor.

Part A of the study is to determine the dose of the study drug. Part A is divided into two sections, A1 and A2. In Part A1, patients will be given study drug without a lead-in period. In Parts A2 and B, patients will have a lead-in period of 2 or 4 weeks with a low dose of LY2784544 prior to taking a higher dose of LY2784544. Part B of the study is to confirm the safety of the dose and schedule.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of polycythemia vera (PV), essential thrombocythemia (ET), or myelofibrosis (MF) as defined by the World Health Organization (WHO) diagnostic criteria for myeloproliferative neoplasms and meet the following additional sub-type specific criteria:

A. PV: has failed or is intolerant of standard therapies or refuses to take standard medications

B. ET: has failed or is intolerant of standard therapies or refuses to take standard medications

C. MF (patients with MF must meet at least one of the following):

i. has intermediate or high-risk MF according to the Lille scoring system; or

ii. has symptomatic MF with spleen greater than 10 cm below left costal margin; or

iii. has post-polycythemic MF; or

iv. has post-ET MF

* Have a quantifiable JAK2 V617F mutation
* Have discontinued all previous approved therapies for myeloproliferative disorders, including any chemotherapy, immunomodulating therapy (for example, thalidomide, interferon-alpha), immunosuppressive therapy (for example, corticosteroids greater than 10 mg/day prednisone or equivalent), radiotherapy, and erythropoietin, thrombopoietin, or granulocyte colony stimulating factor for at least 14 days and recovered from the acute effects of therapy. Hydroxyurea used to control blood cell counts is permitted at study entry if the subject has been maintained on a stable dose for at least 4 weeks. Low-dose acetylsalicylic acid (aspirin) is permitted as well

Exclusion Criteria:

* Have received treatment within 14 days of the initial dose of study drug with an experimental agent that has not received regulatory approval for any indication
* Are currently being treated with agents that are metabolized by CYP3A4 with a narrow therapeutic margin (for example, alfentanil, cyclosporine, diergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus) or CYP2B6 (for example, cyclophosphamide, ifosfamide, tamoxifen, efavirenz, propofol, methadone, and bupropion)
* Are currently being treated with warfarin or one of its derivatives which is known to alter levels of protein C or protein S. An exception to this criterion will be allowed for patients with a prior history of Budd-Chiari Syndrome who are being treated with warfarin or one of its derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Determination of a recommended Phase 2 dosing regimen | Time of first dose until last dose
Number of participants with clinical significant effects | Time of first dose until last dose

SECONDARY OUTCOMES:
Preliminary pharmacokinetics of LY2784544 (Cmax) | Part A1: Day 1,2,15, and 29; Part A2: Day 7, 14, 21, 28, 29, 56, and 57; Part B: Day 1, 29, 57, and 113
Preliminary pharmacokinetics of LY2784544 (AUC) | Part A1: Day 1,2,15, and 29; Part A2: Day 7, 14, 21, 28, 29, 56, and 57; Part B: Day 1, 29, 57, and 113
Malignant clone burden | Part A1: Baseline (2 times), Weeks 13, 21 and every 6 months while patient is on study; Parts A2 and B: Baseline (2 times), Weeks 5, 8, 17, 25 and every 6 months while patient is on study

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah

REFERENCES:
- [Derived] Verstovsek S, Mesa RA, Salama ME, Li L, Pitou C, Nunes FP, Price GL, Giles JL, D'Souza DN, Walgren RA, Prchal JT. A phase 1 study of the Janus kinase 2 (JAK2)V617F inhibitor, gandotinib (LY2784544), in patients with primary myelofibrosis, polycythemia vera, and essential thrombocythemia. Leuk Res. 2017 Oct;61:89-95. doi: 10.1016/j.leukres.2017.08.010. Epub 2017 Aug 31. PMID 28934680